CLINICAL TRIAL: NCT06095102
Title: A Phase 3 Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of JNJ-77242113 for the Treatment of Participants With Plaque Psoriasis Involving Special Areas
Brief Title: A Study of JNJ-77242113 for the Treatment of Participants With Plaque Psoriasis Involving Special Areas (Scalp, Genital, and/or Palms of the Hands and the Soles of the Feet)
Acronym: ICONIC-TOTAL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 77242113PSO3003; 77242113PSO3003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2023-10-18; First posted 2023-10-23 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- JNJ-77242113 (Experimental): Participants will receive JNJ-77242113 from Week 0 through Week 156.
  Interventions: Drug: JNJ-77242113
- Placebo (Placebo Comparator): Participants will receive placebo from Week 0 through Week 16 and thereafter will receive JNJ-77242113 from Week 16 through Week 156.
  Interventions: Drug: JNJ-77242113; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-77242113 — JNJ-77242113 will be administered orally.
Drug: Placebo — Placebo will be administered orally.
  Arms: Placebo

SUMMARY:
The purpose of the study is to see how effective JNJ-77242113 is in participants with plaque psoriasis affecting special areas (scalp, genital, and/or palms of the hands and the soles of the feet).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of plaque psoriasis, with or without psoriatic arthritis (PsA), for at least 26 weeks prior to the first administration of study intervention
* Candidate for phototherapy or systemic treatment for plaque psoriasis
* Need to meet criteria: Total body surface area (BSA) greater than or equal to (>=)1 percent (%) at screening and baseline, and investigator global assessment (IGA) (overall) >=2 at screening and baseline and at least one of the following: scalp-specific investigator global assessment (ss-IGA) score >=3 at screening and baseline, and/or static physician's global assessment of genitalia (sPGA-G) >=3 at screening and baseline, and/or physician's global assessment of hands and feet (hf-PGA) score >=3 at screening and baseline
* Failed to respond to at least 1 topical therapy (example, corticosteroids, calcineurin inhibitors, and/or vitamin D analogs) used for treatment of psoriasis
* Confirmation of plaque psoriasis in a non-special area (example, areas excluding scalp, genital, palmoplantar) at screening and baseline

Exclusion Criteria:

* Nonplaque form of psoriasis (example, erythrodermic, guttate, or pustular)
* Dermatoses other than plaque psoriasis (such as contact dermatitis) or palmoplantar pustulosis of the palmoplantar area (if hf-PGA >=3 at baseline)
* Current drug-induced psoriasis (example, a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium)
* A current diagnosis or signs or symptoms of severe, progressive, or uncontrolled renal, liver, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Known allergies, hypersensitivity, or intolerance to JNJ-77242113 or its excipients

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2027-02-17 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving an Investigator's Global Assessment (IGA) Score of 0 or 1 and Greater Than or Equal to (>=) 2 Grade Improvement From Baseline at Week 16 | Baseline and Week 16
  Percentage of participants who achieve an IGA score of 0 or 1 and >=2 grade improvement from baseline at Week 16 will be reported. The IGA documents the investigator's assessment of the participants psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).

SECONDARY OUTCOMES:
Percentage of Participants Achieving Scalp-specific Investigator Global Assessment (ss-IGA) Score of 0 or 1 at Week 16 | Week 16
  Percentage of participants achieving ss-IGA score of 0 or 1 at Week 16 will be reported. The ss-IGA instrument is used to evaluate the disease severity of scalp psoriasis. The lesions are assessed in terms of the clinical signs of redness, thickness, and scaliness which are scored as: absence of disease (0), very mild disease (1), mild disease (2), moderate disease (3), and severe disease (4).
Percentage of Participants Achieving Psoriasis Scalp Severity Index (PSSI) 90 at Week 16 | Baseline and Week 16
  Percentage of participants achieving PSSI 90 (90% reduction in PSSI score from baseline) at Week 16 will be reported. The PSSI is a scalp-specific modification of the PASI based on the extent of involvement and the severity of erythema, infiltration, and desquamation. Involvement and severity of psoriasis on the PSSI is scored by physicians on a scale from 0 to 72, where 0 = no psoriasis and higher scores indicate more severe disease.
Percentage of Participants Achieving a Static Physician's Global Assessment of Genitalia (sPGA-G) Score of 0 or 1 at Week 16 | Week 16
  Percentage of participants achieving a sPGA-G Score of 0 or 1 at Week 16 will be reported. The sPGA-G is a 6-point scale to assess the severity of genital psoriasis at a given time point. The sPGA-G evaluates erythema, plaque elevation, and scale of genital psoriatic lesions. The severity of genital psoriasis is assessed as clear (0), minimal (1), mild (2), moderate (3), severe (4), and very severe (5).
Percentage of Participants Achieving a Physician's Global Assessment of Hands and Feet (hf-PGA) Score of 0 or 1 at Week 16 | Week 16
  Percentage of participants achieving a hf-PGA score of 0 or 1 at Week 16 will be reported. The hf-PGA assesses the severity of hand and foot psoriasis using a 5-point scale to score the plaques on the hands and feet as: clear (0), almost clear (1), mild (2), moderate (3), and severe (4).
Percentage of Participants Achieving Psoriasis Symptom and Sign Diary (PSSD) Symptoms Score of 0 at Week 16 | Week 16
  Percentage of participants achieving PSSD symptoms score of 0 at Week 16 will be reported. The PSSD includes patient-reported outcome (PRO) questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Percentage of Participants Achieving >=4 Point Improvement From Baseline in PSSD Itch Score at Week 16 | Baseline and Week 16
  Percentage of participants achieving >=4 Point improvement from baseline in PSSD itch score at Week 16 will be reported. The PSSD includes PRO questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Percentage of Participants Achieving Genital Psoriasis Sexual Frequency Questionnaire (GenPs-SFQ) Item 2 score of 0 or 1 at Week 16 | Week 16
  Percentage of participants achieving GenPs-SFQ item 2 score of 0 or 1 at Week 16 will be reported. The GenPs-SFQ is a 2-item participant-reported instrument used to assess the impact of genital psoriasis on the frequency of sexual activity in the last 7 days. Item 1 assesses overall frequency of sexual activity in the last 7 days (none/zero, once, or 2 or more times), and item 2 assesses how frequently genital psoriasis symptoms have limited the frequency of sexual activity in the last 7 days (never [0], rarely [1], sometimes [2], often [3], or always [4]).
Percentage of Participants Achieving >=4-Point Improvement From Baseline in Scalp Itch Numeric Rating Scale (NRS) Score at Week 16 | Baseline and Week 16
  Percentage of participants achieving >=4-point improvement from baseline in scalp itch NRS score at Week 16 will be reported. The Scalp Itch NRS is a single item instrument that evaluates the severity of scalp itch in adult and adolescent populations over the past 24 hours. The instrument uses an NRS score ranging from 0 (no scalp itch) to 10 (worst scalp itch imaginable).
Percentage of Participants Achieving >=4-Point Improvement From Baseline in Genital Psoriasis Symptoms Scale (GPSS) Genital Itch NRS Score at Week 16 | Baseline and Week 16
  Percentage of participants achieving >=4-point improvement from baseline in GPSS genital itch NRS score at Week 16 will be reported. The GPSS is a participant-administered assessment of 8 symptoms: itch, pain, discomfort, stinging, burning, redness, scaling, and cracking. Each respondent is asked to answer the questions based on the psoriasis symptoms in his or her genital area. The overall severity for each individual genital psoriasis symptom is indicated by selecting the number from an NRS of 0 to 10 that best describes the worst level of each symptom in the genital area in the past 24 hours, ranging from 0 (no severity) to 10 (worst imaginable severity).
Number of Participants with Adverse Events (AEs) | Up to 165 weeks
  An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Number of Participants with Serious Adverse Events (SAEs) | Up to 165 weeks
  An SAE is any AE which results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product, or is medically important.
Percentage of Participants Achieving Psoriasis Area and Severity Index (PASI) 90 Response at Week 16 | Baseline and Week 16
  Percentage of participants achieving PASI 90 response (>=90% improvement in PASI from baseline) at Week 16 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Percentage of Participants Achieving PASI 75 Response at Week 16 | Baseline and Week 16
  Percentage of participants achieving PASI 75 response (>=75% improvement in PASI from baseline) at Week 16 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Change from Baseline in PASI Total Score at Week 16 | Baseline and Week 16
  Change from baseline in PASI total score at Week 16 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: head, trunk, upper, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 (none) to 4 (severe). The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Change From Baseline in BSA at Week 16 | Baseline and Week 16
  Change from baseline in BSA at Week 16 will be reported. BSA is a commonly used measure of extent of skin disease. It is defined as the percentage of surface area of the body involved with the condition being assessed (that is, plaque psoriasis).
Percent Change From Baseline in Modified Nail Psoriasis Areas and Severity Index (mNAPSI) Score at Week 16 | Baseline and Week 16
  Percent change from baseline in mNAPSI Score at Week 16 will be reported. The mNAPSI is an index used for assessing and grading the severity of nail psoriasis. Each of the participant's ten fingernails are evaluated on 7 features. The first three features are each scored from 0 to 3 in severity and are (1) onycholysis and oil-drop dyschromia, (2) pitting, and (3) nail plate crumbling. The next four features are each scored 0 -absent or 1 -present, and are (1) leukonychia, (2) splinter hemorrhages, (3) nail bed hyperkeratosis, and (4) red spots in the lunula. The score ranges from 0-13 per nail, and 0-130 for all fingernails.
Percentage of Participants Achieving Fingernail Physician's Global Assessment (f-PGA) Score of 0 or 1 at Week 16 | Week 16
  Percentage of participants achieving f-PGA score of 0 or 1 at Week 16 will be reported. The f-PGA is used to evaluate the current status of a participant's fingernail psoriasis on a scale of 0 to 4 similar (clear [0], minimal [1], mild [2], moderate [3], or severe [4]). Higher score indicated severe disease.
Percentage of Participants Achieving an IGA Score of 0 at Week 16 | Week 16
  Percentage of participants achieving an IGA Score of 0 at Week 16 will be reported. The IGA documents the investigator's assessment of the participants psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Percentage of Participants Achieving PSSD Symptom Score of 0 at Week 8 | Week 8
  Percentage of participants achieving PSSD symptom score of 0 at Week 8 will be reported. The PSSD includes PRO questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Change From Baseline in PSSD Symptom Score at Week 16 | Baseline and Week 16
  Change from baseline in PSSD symptom score at Week 16 will be reported. The PSSD includes PRO questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Percentage of Participants Achieving >=4-Point Improvement From Baseline in PSSD Itch Score at Week 4 | Baseline and Week 4
  Percentage of participants achieving >=4-point improvement from baseline in PSSD itch score at Week 4 will be reported. The PSSD includes PRO questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Change From Baseline in PSSD Sign Score at Week 16 | Baseline and Week 16
  Change from baseline in PSSD sign score at Week 16 will be reported. The PSSD includes PRO questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Percentage of Participants Achieving PSSD Sign Score of 0 at Week 16 | Week 16
  Percentage of participants achieving PSSD sign score of 0 at Week 16 will be reported. The PSSD includes PRO questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Percentage of Participants Achieving Dermatology Life Quality Index (DLQI) Score of 0 or 1 at Week 16 | Week 16
  Percentage of participants achieving DLQI score of 0 or 1 at Week 16 will be reported. The DLQI is a dermatology specific health-related quality of life (HRQoL) instrument designed to assess the impact of the disease on a participant's HRQoL. It is a 10-item questionnaire that assesses HRQoL over the past week and in addition to evaluating overall HRQoL, can be used to assess 6 different aspects that may affect quality of life: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. The total score ranges from 0 to 30 with a higher score indicating greater impact on HRQoL.
Percentage of Participants Achieving Children's Dermatology Life Quality Index (CDLQI) score of 0 or 1 at Week 16 | Week 16
  Percentage of participants achieving CDLQI score of 0 or 1 at Week 16 will be reported. The CDLQI is a dermatology-specific quality of life (QoL) instrument designed to assess the impact of the disease on a child's QoL. The CDLQI, a 10-item questionnaire has 4-item response options and a recall period of 1 week. The CDLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0; the higher the score, the greater the impairment in QoL.
Change From Baseline in Domain Scores of the Patient-reported Outcomes Measurement Information System-29 (PROMIS-29) Score at Week 16 | Baseline and Week 16
  Change from baseline in PROMIS-29 domain scores at week 16 will be reported. The PROMIS-29 is a 29-item generic HRQoL instrument assessing 7 PROMIS domains (depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social roles and activities) with 4 questions for each domain. These questions are ranked on a 5-point Likert scale. There is also a numerical rating scale that ranges from 0 (No pain) to 10 (Worst pain imaginable) for pain intensity. The raw domain scores are converted to standardized T-scores with a mean of 50 and a standard deviation of 10. Higher scores on anxiety, depression, fatigue, sleep disturbance, and pain interference indicate more severe symptoms. Higher scores on physical function and social participation indicate better health outcomes.
Change From Baseline in Domain Scores of the Patient-reported Outcomes Measurement Information System-25 (PROMIS-25) Score at Week 16 | Baseline and Week 16
  Change from baseline in domain scores of the PROMIS-25 score at Week 16 will be reported. The PROMIS-25 will be utilized in the adolescent population and is a 25-item generic HRQoL survey. Six PROMIS domains (physical function mobility, anxiety, depressive symptoms, fatigue, peer relationships, pain interference) are each assessed with 4 questions. There is also one 11-point rating scale for pain intensity. The instrument is designed for use in ages 8-17 years of age and can be self-administered.
Change From Baseline in Palmoplantar Quality of Life Instrument (ppQLI) Score at Week 16 | Baseline and Week 16
  Change from baseline in ppQLI score at Week 16 will be reported. The ppQLI assesses impact on patient quality of life due to palmoplantar psoriasis over the past month in adult and adolescent populations. Fifteen items evaluate hand functionality, pain, and social impact due to psoriasis. Fourteen items evaluate foot functionality, pain, and physical limitations due to psoriasis. All items use verbal rating scales ranging from 1 to 5. The ppQLI yields a score for hands, ranging from 15 to 80, and a score for feet, ranging from 14 to 70.
Change From Baseline in Genital Psoriasis Symptoms Scale (GPSS) Total Score at Week 16 | Baseline and Week 16
  Change from baseline in GPSS total score at Week 16 will be reported. The GPSS is a participant-administered assessment of 8 symptoms: itch, pain, discomfort, stinging, burning, redness, scaling, and cracking. Each respondent is asked to answer the questions based on the psoriasis symptoms in his or her genital area. The overall severity for each individual genital psoriasis symptom is indicated by selecting the number from an NRS of 0 to 10 that best describes the worst level of each symptom in the genital area in the past 24 hours, ranging from 0 (no severity) to 10 (worst imaginable severity).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research &Development, LLC Clinical trial, Study Director — Janssen Research & Development, LLC
Locations (90):
- United States (28):
  - Center for Dermatology and Plastic Surgery, Scottsdale, Arizona
  - Johnson Dermatology, Fort Smith, Arkansas
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Forcare Clinical Research Inc, Tampa, Florida
  - Hamilton Research LLC, Alpharetta, Georgia
  - Arlington Dermatology, Rolling Meadows, Illinois
  - Dundee Dermatology, West Dundee, Illinois
  - Dawes Fretzin Clinical Research Group LLC, Indianapolis, Indiana
  - Indiana Clinical Trial Center, Plainfield, Indiana
  - Dermatology and Advanced Aesthetics, Lake Charles, Louisiana
  - Allcutis Research, Beverly, Massachusetts
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Skin Specialists, Omaha, Nebraska
  - Schweiger Dermatology Group, East Windsor, New Jersey
  - Optima Research, Boardman, Ohio
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Paddington Testing Co, Inc., Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Arlington Research Center, Inc., Arlington, Texas
  - Center for Clinical Studies, Houston, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
  - Cope Family Medicine - Ogden Clinic, Bountiful, Utah
  - Frontier Derm Partners CRO, LLC, Mill Creek, Washington
- Argentina (4):
  - CIPREC, Buenos Aires
  - Centro Privado de Medicina Familiar, Buenos Aires
  - Conexa Investigacion Clinica S.A., CABA
  - CEDIC Centro de Investigacion clinica, Caba
- Canada (7):
  - Alberta DermaSurgery Centre, Edmonton, Alberta
  - Lynderm Research Inc., Markham, Ontario
  - Skin Centre for Dermatology, Peterborough, Ontario
  - York Dermatology Clinic and Research Centre, Richmond Hill, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Centre De Recherche Dermatologique Du Quebec Metropolitain, Québec, Quebec
  - Skinsense Medical Research, Saskatoon, Saskatchewan
- Germany (9):
  - ISA - Interdisciplinary Study Association GmbH, Berlin
  - CRS Clinical Research Services Berlin GmbH, Berlin
  - Niesmann & Othlinghaus GbR, Bochum
  - Rosenpark Research GmbH, Darmstadt
  - Medizinische Fakultaet Carl Gustav Carus Technische Universitaet Dresden, Dresden
  - Universitaetsklinikum Frankfurt, Frankfurt am Main
  - Dermatologikum Hamburg Gmbh, Hamburg
  - Klinische Forschung Schwerin GmbH, Schwerin
  - Hautarztpraxis, Witten
- Hungary (6):
  - Pecsi Tudomanyegyetem, Borgyogyaszati Klinika
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Derma-B Kft, Debrecen
  - SZTE AOK Szent-Gyorgyi Albert Klinikai Kozpont, Borgyogyaszati és Allergologiai Klinika, Szeged
  - Allergo-Derm Bakos Kft., Szolnok
  - Medmare Egeszsegugyi Es Szolgaltato Bt., Veszprém
- Poland (13):
  - Osteo-Medic s.c A. Racewicz, J Supronik, Bialystok
  - Specderm Poznanska sp j, Bialystok
  - Centrum Medyczne dr Rajzer Sp z o o, Krakow
  - Specjalistyczny gabinet dermatologiczny Aplikacyjno Badawczy Marek Brzewski Pawel Brzewski Spolka Cywilna, Krakow
  - Centrum Medyczne Promed, Krakow
  - Dermed Centrum Medyczne Sp z o o, Lodz
  - Dermodent Centrum Medyczne Aldona Czajkowska Rafal Czajkowski S C, Osielsko
  - SOLUMED Centrum Medyczne, Poznan
  - Clinical Research Center sp z o o MEDIC R s k, Poznan
  - Dorota Bystrzanowska High-Med. Przychodnia Specjalistyczna, Warsaw
  - Klinika Ambroziak Dermatologia, Warsaw
  - Wro Medica, Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
- South Korea (5):
  - Pusan National University Hospital, Busan
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (8):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp. Del Mar, Barcelona
  - Hosp. Sant Joan de Deu, Esplugues de Llobregat
  - Hosp. Univ. San Cecilio, Granada
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. de Manises, Manises
  - Hosp. Virgen Macarena, Seville
  - Hosp. Univ. I Politecni La Fe, Valencia
- Taiwan (4):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - National Taiwan University Hospital Hsin Chu Branch, Taoyuan District
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Turkey (Türkiye) (3):
  - Necmettin Erbakan University Meram Medical Faculty, Konya
  - Ondokuz Mayis University, Samsun
  - Karadeniz Teknik University Medical Faculty, Trabzon
- United Kingdom (3):
  - London North West University Healthcare NHS Trust, Harrow
  - Salford Royal Hospital, Salford
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Gooderham M, Lain E, Bissonnette R, Huang YH, Lynde CW, Hoffmann M, Song EJ, Weirich O, Ceitlin RHG, Rubens JH, DeLozier AM, Ota T, Hsu MC, Li S, DeKlotz CMC, Nunes F, Warren RB. Targeted Oral Peptide Icotrokinra for Psoriasis Involving High-Impact Sites. NEJM Evid. 2025 Dec;4(12):EVIDoa2500155. doi: 10.1056/EVIDoa2500155. Epub 2025 Nov 5. PMID 41191932